CLINICAL TRIAL: NCT00570934
Title: Effect of Supplementation With 2000 International Units (IU) Vitamin D, 1gm Calcium or Both on Calcium Absorption and Bone Mineralization in Children With Juvenile Rheumatoid Arthritis
Brief Title: Supplementation With Vitamin D, Calcium or Both on Calcium Absorption and Bone Mineral Content in Children With JRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5387
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): order of interventions placebo,calcium, cholecalciferol, calcium plus cholecalciferol
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: Calcium; Dietary Supplement: Calcium and cholecalciferol; Drug: Placebo
- Calcium (Experimental): order of treatment calcium, placebo, calcium plus cholecalciferol, cholecalciferol
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: Calcium; Dietary Supplement: Calcium and cholecalciferol; Drug: Placebo
- Cholecalciferol (Experimental): order of treatments cholecalciferol, calcium and Cholecalciferol, placebo, and calcium
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: Calcium; Dietary Supplement: Calcium and cholecalciferol; Drug: Placebo
- Calcium and cholecalciferol (Experimental): order of treatment calcium and cholecalciferol, cholecalciferol, calcium, placebo
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: Calcium; Dietary Supplement: Calcium and cholecalciferol; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 2000IU Cholecalciferol P.O. Q.D.
Dietary Supplement: Calcium — 1 gm calcium as calcium carbonate
Dietary Supplement: Calcium and cholecalciferol — 2000IU cholecalciferol and 1 gm calcium P.O. Q.D. for 6 months
Drug: Placebo — Placebo

SUMMARY:
2000 international units (IU) vitamin D, 1 gram (gm) calcium, or both given to children with Juvenile Rheumatoid Arthritis (JRA) may increase percent true calcium absorption, bone mineral turnover and/or bone mineralization.

DETAILED DESCRIPTION:
Supplementation With 2000 IU Vitamin D, 1 gm Calcium or Both on Calcium Absorption and Bone Mineralization in Children With Juvenile Rheumatoid Arthritis may increase percent true calcium absorption, bone mineral turnover and/or bone mineralization.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Rheumatoid arthritis

Exclusion Criteria:

* Steroid use

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 1995-03; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Percent true calcium absorption | After 6 months of treatment

SECONDARY OUTCOMES:
Bone Mineralization by Dual Energy x-ray absorption | After 6 months treatment plus 3 month washout

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Hillman, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospitals and clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillman LS, Cassidy JT, Chanetsa F, Hewett JE, Higgins BJ, Robertson JD. Percent true calcium absorption, mineral metabolism, and bone mass in children with arthritis: effect of supplementation with vitamin D3 and calcium. Arthritis Rheum. 2008 Oct;58(10):3255-63. doi: 10.1002/art.23809. PMID 18821668